CLINICAL TRIAL: NCT06883136
Title: Efficacy and Safety of Sintilimab Combined with Platinum-containing Double-agent Chemotherapy in First-line Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer in Elderly Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Degan Lu, prof., Qianfoshan Hospital
Other Study IDs: YXLL-KY-2024(127)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Sintilimab; Non-Small Cell Lung Cancer; Elderly population
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; Gemcitabine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sintilimab in combination with chemotherapy containing platinum
  Interventions: Drug: Sintilimab+Cis-platinum/Carboplatin with Pemetrexed or Gemcitabine

INTERVENTIONS:
Drug: Sintilimab+Cis-platinum/Carboplatin with Pemetrexed or Gemcitabine — 1. Sintilimab, 200mg, intravenous infusion on day 1 of each cycle, every 3 weeks as a cycle (Q3W), until disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor therapy, or termination of treatment for other reasons specified in the protocol; The longest treatment time of sintilimab was 24 months.
  2. Chemotherapy regimen:
  1) Pemetrexed combined with platinum regimen (non-squamous cell carcinoma) : pemetrexed 500mg/m2, intravenous infusion on day 1 of each cycle, cisplatin 75mg/m2 or carboplatin AUC 5, intravenous infusion on day 1 of each cycle, every 3 weeks (Q3W) for a total of 4-6 cycles.
  2) Gemcitabine plus platinum regimen (squamous cell carcinoma) : gemcitabine 1000mg/m2 intravenously on days 1 and 8 of each cycle, cisplatin 75mg/m2 or carboplatin: AUC 5, intravenous infusion on day 1 of each cycle, every 3 weeks (Q3W) for 4-6 cycles.

SUMMARY:
To investigate the efficacy and safety of sindilizumab combined with platinum-containing dual chemotherapy in first-line treatment of elderly patients with locally advanced or metastatic non-small cell lung cancer (NSCLC).

This study was an observational, prospective, single-arm, single-center study. Specific dosing regimens are as follows:

1. Sintilimab, 200mg, intravenous infusion on day 1 of each cycle, every 3 weeks as a cycle (Q3W), until disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor therapy, or termination of treatment for other reasons specified in the protocol; The longest treatment time of sintilimab was 24 months.
2. Chemotherapy regimen:

1) Pemetrexed combined with platinum regimen (non-squamous cell carcinoma) : pemetrexed 500mg/m2, intravenous infusion on day 1 of each cycle, cisplatin 75mg/m2 or carboplatin AUC 5, intravenous infusion on day 1 of each cycle, every 3 weeks (Q3W) for a total of 4-6 cycles. Participants who did not progress after 4 to 6 cycles received maintenance pemetrexed monotherapy at the same dose and cycle as before until disease progression, death, unacceptable toxicity, withdrawal of consent, initiation of a new antineoplastic therapy, or discontinuation for other protocol-specified reasons.

2) Gemcitabine plus platinum regimen (squamous cell carcinoma) : gemcitabine 1000mg/m2 intravenously on days 1 and 8 of each cycle, cisplatin 75mg/m2 or carboplatin: AUC 5, intravenous infusion on day 1 of each cycle, every 3 weeks (Q3W) for 4-6 cycles. Participants who did not progress after 4 to 6 cycles received maintenance gemcitabine monotherapy at the same dose and cycle as before until disease progression, death, unacceptable toxicity, withdrawal of consent, initiation of a new antineoplastic therapy, or discontinuation for other protocol-specified reasons.

Patients are assessed for measurable disease at baseline, 6 weeks, 12 weeks after starting treatment, and every 9 weeks thereafter according to RECIST 1.1 criteria during the treatment period until disease progression or intolerable toxicity withdrawal. Following discontinuation of treatment, subjects are followed for survival status every 3 months until death. Subject safety was assessed during treatment according to NCI CTCAE Version 5.0 criteria. Subjects who experience an AE should be followed until the AE returns to baseline.

DETAILED DESCRIPTION:
To investigate the efficacy and safety of sindilizumab combined with platinum-containing dual chemotherapy in first-line treatment of elderly patients with locally advanced or metastatic non-small cell lung cancer (NSCLC).

This study was an observational, prospective, single-arm, single-center study. Specific dosing regimens are as follows:

1. Sintilimab, 200mg, intravenous infusion on day 1 of each cycle, every 3 weeks as a cycle (Q3W), until disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor therapy, or termination of treatment for other reasons specified in the protocol; The longest treatment time of sintilimab was 24 months.
2. Chemotherapy regimen:

1) Pemetrexed combined with platinum regimen (non-squamous cell carcinoma) : pemetrexed 500mg/m2, intravenous infusion on day 1 of each cycle, cisplatin 75mg/m2 or carboplatin AUC 5, intravenous infusion on day 1 of each cycle, every 3 weeks (Q3W) for a total of 4-6 cycles. Participants who did not progress after 4 to 6 cycles received maintenance pemetrexed monotherapy at the same dose and cycle as before until disease progression, death, unacceptable toxicity, withdrawal of consent, initiation of a new antineoplastic therapy, or discontinuation for other protocol-specified reasons.

2) Gemcitabine plus platinum regimen (squamous cell carcinoma) : gemcitabine 1000mg/m2 intravenously on days 1 and 8 of each cycle, cisplatin 75mg/m2 or carboplatin: AUC 5, intravenous infusion on day 1 of each cycle, every 3 weeks (Q3W) for 4-6 cycles. Participants who did not progress after 4 to 6 cycles received maintenance gemcitabine monotherapy at the same dose and cycle as before until disease progression, death, unacceptable toxicity, withdrawal of consent, initiation of a new antineoplastic therapy, or discontinuation for other protocol-specified reasons.

Patients are assessed for measurable disease at baseline, 6 weeks, 12 weeks after starting treatment, and every 9 weeks thereafter according to RECIST 1.1 criteria during the treatment period until disease progression or intolerable toxicity withdrawal. Following discontinuation of treatment, subjects are followed for survival status every 3 months until death. Subject safety was assessed during treatment according to NCI CTCAE Version 5.0 criteria. Subjects who experience an AE should be followed until the AE returns to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent before performing any trial-related procedures;
2. Age 60-80 years old;
3. Study participants with histologically or cytologically confirmed locally advanced (IIIB-IIIC) or metastatic (stage IV) NSCLC (International Association for the Study of Lung Cancer and American Joint Committee on Classification of Cancer 8th Edition TNM stage), inoperable and definitive concurrent chemoradiotherapy without previous systemic therapy;
4. No EGFR gene sensitive mutation or ALK gene fusion mutation was confirmed by histological specimens; At least one radiographic measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.

6. Had not received any previous systemic antitumor therapy for advanced/metastatic disease. Participants who had received previous platinum-based adjuvant/neoadjuvant chemotherapy or definitive chemoradiotherapy for advanced disease were allowed if they had disease progression or relapse at least 6 months after the last dose of chemotherapy.

7. Study participants with asymptomatic or symptomatic stable brain metastases after local treatment were allowed to enroll as long as the study participant met the following conditions:

1) measurable lesions outside the central nervous system 2) no central nervous system symptoms or worsening of symptoms for at least 2 weeks 3) no glucocorticoid treatment was required, glucocorticoid treatment was discontinued within 7 days before the first dose, or the glucocorticoid dose was stable and reduced to less than 10mg/ day prednisone (or equivalent) within 7 days before the first dose 8. Study participants were allowed to receive palliative radiation therapy 7 days before the first dose of study drug and with a return of radiotherapy-related toxicity to grade 1 or less (CTCAE5.0); 9.ECOG score 0-2; 10. Expected survival time >3 months; 11. Adequate organ function, study participants had to meet the following laboratory measures:

1. absolute neutrophil count (ANC) ≥1.5x109/L without using granulocyte colony-stimulating factor for the past 14 days;
2. platelet count ≥100×109/L without blood transfusion in the past 14 days;
3. hemoglobin >9g/dL in the absence of blood transfusion or erythropoietin use in the past 14 days;
4. Total bilirubin ≤1.5 times upper limit of normal value (ULN)
5. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤2.5 ×ULN (participants with liver metastases were allowed ALT or AST ≤5×ULN);
6. serum creatinine ≤1.5 times ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
7. good coagulation function, defined as INR or PT ≤1.5 times ULN;
8. Euthyroid, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH level was outside the normal range, participants were eligible if their total T3 (or FT3) and FT4 levels were within the normal range.
9. Myocardial enzymes within the normal range (isolated laboratory abnormalities that were judged by the investigators as not clinically significant were also allowed).

12. Study participants were discretionary in applying the study regimen.

Exclusion Criteria:

1. Malignant diseases other than NSCLC diagnosed within 5 years before the first dose (excluding radical skin basal cell carcinoma, skin squamous cell carcinoma, and/or radical resection in situ carcinoma);
2. Are currently participating in an interventional clinical study treatment, or have received another study drug or study device within 4 weeks before the first dose;
3. Prior therapy with: Anti-pd-1, anti-PD-L1 agents or agents targeting another T-cell receptor that stimulates or coinhibits it (e.g., CTLA-4, OX-40, CD137) Such as tislelizumab, toripalimab, carrelizumab, atezolizumab, slulizumab, pembrolizumab, paiampalimab, nivolumab, duvalumab, ipilimumab, etc.
4. Received systemic treatment with Chinese patent medicine or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use to control pleural effusion) with indications for anti-NSCLC within 2 weeks before the first dose;
5. Active autoimmune disease requiring systemic therapy (e.g., disease-modifying agents, glucocorticoids, or immunosuppressive agents) occurred within 2 years before the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) were not considered systemic therapy;
6. Presence of clinically uncontrollable pleural/peritoneal effusion (participants who did not require fluid drainage or who stopped drainage for 3 days without a significant increase in fluid volume were eligible);
7. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
8. Patients with known allergy to sintilimab, pemetrexed, gemcitabine, carboplatin, cisplatin and other active ingredients or excipients of the study drug;
9. Has not fully recovered from any intervention-related toxicity and/or complications before starting treatment (i.e., grade ≤1 or baseline, excluding fatigue or alopecia);
10. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive);
11. Untreated active hepatitis B (defined as both HBsAg positivity and HBV-DNA copies greater than the upper limit of normal in the laboratory at the participating center);

Note: Hepatitis B study participants were eligible if they met the following criteria:

1. HBV viral load <1000 copies /ml (200 IU/ml) before the first dose, study participants should receive anti-HBV therapy throughout the study chemotherapy to avoid viral reactivation
2. Study participants with anti-HBc (+), HBsAg (-), anti-hbs (-), and HBV viral load (-) do not require prophylactic anti-HBV therapy, but close monitoring for viral reactivation is required 12. Active HCV-infected study participants with positive HCV antibodies and HCV-RNA levels above the lower limit of detection; 13. A live vaccine dose within 30 days before the first dose (cycle 1, day 1); Note: Administration of injectable inactivated virus vaccine against seasonal influenza within 30 days before the first dose is allowed; Live, attenuated, intranasal influenza vaccine was not allowed.

14. The presence of any serious or uncontrolled systemic illness, such as:

1. significant rhythm, conduction or morphological abnormalities in resting ECG, such as complete left bundle branch block, ≥ Ⅱ degree heart block, ventricular arrhythmia or atrial fibrillation;
2. unstable angina, congestive heart failure, New York Heart Association (NYHA) grade ≥ 2 chronic heart failure;
3. myocardial infarction within 6 months before enrollment;
4. poor blood pressure control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
5. patients had a history of noninfectious pneumonia requiring glucocorticoid treatment within 1 year before the first dose of glucocorticoid, or current clinically active interstitial lung disease;
6. active pulmonary tuberculosis;
7. presence of active or uncontrolled infection requiring systemic therapy;
8. presence of clinically active diverticulitis, abdominal abscess, or gastrointestinal obstruction;
9. liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
10. poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L);
11. Urine routine test showed urinary protein ≥++ and confirmed 24-hour urinary protein quantitation > 1.0 g;
12. participants with a psychiatric disorder who were unable to cooperate with treatment; Any medical history or evidence of illness, abnormal treatment or laboratory values, or other conditions that might interfere with the results of the trial or prevent full participation in the study were considered by the investigators to be other potential risks that might preclude participation.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants with histologically or cytologically confirmed, locally advanced or metastatic (stage IIIB, IIIC, IV) NSCLC that was inoperable and not amenable to definitive concurrent chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-03-12 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-06-29 (Estimated)

PRIMARY OUTCOMES:
ORR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months]
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Progression-free survival
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  overall survival
DCR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Disease Control Rate
DoR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Duration of Response,

CONTACTS AND LOCATIONS:
Overall Officials: Min Gao, Study Chair — Qianfoshan Hospital
Locations (2):
- China (2):
  - Degan Lu, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided